CLINICAL TRIAL: NCT07033689
Title: Open-label, Non-randomized, Single-center Study Investigating the Feasibility, Safety, Tolerability and Efficacy of Suizenji in Unresectable Pancreatic Ductal Adenocarcinoma Patients
Brief Title: Feasibility Study of Suizenji, in Patients With Unresectable Pancreatic Ductal Adenocarcinoma (SUNRISE-II)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: SONIRE Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: Sonire-PAC-002
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer,; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Suizenji (an ultrasound-guided HIFU therapy system)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Suizenji (an ultrasound-guided HIFU therapy system) (Experimental): Suizenji (an ultrasound-guided HIFU therapy system)
  Interventions: Device: Suizenji (an ultrasound-guided HIFU therapy system); Drug: Nal-IRI/FL; Drug: mFOLFIRINOX adjuvant chemotherapy; Drug: Gem/nab-PTX

INTERVENTIONS:
Device: Suizenji (an ultrasound-guided HIFU therapy system) — Suizenji (an ultrasound-guided HIFU therapy system)
  Other Names: ultrasound-guided HIFU therapy system
Drug: Nal-IRI/FL — Standard of care
Drug: mFOLFIRINOX adjuvant chemotherapy — standard of care
Drug: Gem/nab-PTX — standard of care

SUMMARY:
This is a feasibility, safety, tolerability, and efficacy research study of an investigational device called "Suizenji", an ultrasound-guided high-intensity focused ultrasound (HIFU) therapy system for the treatment of unresectable pancreatic ductal adenocarcinoma. Focused ultrasound therapy uses a number of small ultrasound generators attached to a bowl-shaped ultrasound generator to emit ultrasound waves from outside to inside the body and focus them on a single point where cancerous cells in the pancreas are located. The targeted area is then heated, which kills the pancreatic cancer cells, and as a result, the patient's life may be prolonged. Experience with Suizenji for pancreatic cancer patients has shown that the "heating" is only a warm feeling in the abdomen during the treatment.

DETAILED DESCRIPTION:
Study Title An Open-label, Non-randomized, Single-center Study Investigating the Feasibility, Safety, Tolerability and Efficacy of Suizenji, an Ultrasound-guided HIFU Therapy System, in Patients with Unresectable Pancreatic Ductal Adenocarcinoma (SUNRISE-II) Objectives Primary objectives

1. To evaluate the safety and tolerability of Suizenji. Secondary objectives
2. To evaluate the overall performance of Suizenji.
3. To explore technical success and preliminary clinical efficacy of Suizenji. Trial Stages Feasibility study Investigational site Stanford Cancer Institute Study Design This is an open-label, non-randomized, single-center study.

The study will consist of:

* A screening period
* HIFU treatment procedure(s) and post-HIFU assessments
* Initiation of 1st line chemotherapy
* Follow-up visits at Month 1 and Month 3
* Long-term follow-up visits until death or up to 5 years Subjects will sign a consent form prior to any study related procedure and will complete baseline screening assessments.

All eligible subjects will be enrolled in the study and will receive HIFU treatment on Day 1. An additional session will be required prior to the initiation of chemotherapy if one of the following; (1) ablation is not completed as planned, or (2) insufficiently ablated per PI's discretion.

After the post HIFU assessment is completed, standard 1st line chemotherapy (FOLFIRINOX (or modified FOLFIRINOX), Gem/nab-PTX, or NALIRIFOX) will be started. The interval from enrollment and the initiation of chemotherapy will be within 2 weeks. All HIFU treatment(s) and post HIFU assessment need to be completed during this 2-week interval.

Subjects will come back for follow-up visits at Month 1 and Month 3. After 3 subjects have completed the one-month evaluation, the DSMB will review the safety and efficacy (except immune response) data up to the Month 1 visit to recommend if the study can continue or if a protocol amendment will be required.

Total 10 subjects are planned to be enrolled. Duration of Subject Participation Subjects will be in the study for up to 3.5 months+ additional long-term follow-up until death or up to 5 years.

Screening: up to 7 days Treatment: 1 day for 1 session + additional sessions if required Follow-up: 3 months Long-term follow-up: until death or up to 5 years Study Population Subjects with unresectable locally advanced or metastatic PDAC.

Inclusion criteria

1. Signed an Institutional Review Board (IRB) approved informed consent document.
2. Men and women ≥ 22 years of age.
3. Histologically or cytologically diagnosed PDAC.
4. Newly diagnosed unresectable*, locally advanced or metastatic disease.
5. Primary tumor accessible to HIFU treatment and visualized on transabdominal ultrasonography.
6. Primary tumor site must be a measurable lesion according to RECIST version 1.1 at baseline.
7. ECOG Performance Status (ECOG-PS) of 0 - 1.
8. Life expectancy ≥ 3 months.
9. Adequate organ function defined by:

   * Neutrophil count: ≥ 1,500/mm3
   * Platelet count: ≥ 50,000/mm3
   * Hemoglobin: ≥ 8.0 g/dl
   * Cr: ≤ 1.7 mg/dl
   * AST, ALT: ≤ 3 x upper limit of normal
   * T-Bil: ≤ 2 x upper limit of normal

Exclusion criteria

1. Subjects with any cancers other than PDAC who are on active treatment.
2. Subjects who had any prior chemotherapy or interventions for PDAC.
3. Obstructive jaundice (except for subjects who have a bile duct stent placed for obstructive jaundice prior to initiation of HIFU treatment).
4. Tumor embolization in the veins surrounding the pancreas.
5. Cysts outside of primary pancreatic tumor which may obstruct the HIFU sonication pathway. However, if the cyst is completely surrounded by pancreatic tumor, the subject can be included.
6. Subjects with > 50% reduction in caliber of the principal hepatic artery and occlusion of the portal vein seen on preoperative screening CT or MRI scan.
7. Allergy to contrast agents (except when manageable by prophylactic steroid).
8. Subjects having a cardiac pacemaker.
9. Congestive heart failure, symptomatic coronary artery disease, arrhythmia poorly controlled by drugs, history of myocardial infarction or unstable angina within the past 6 months.
10. Subjects with peritoneal dissemination.
11. Active infections requiring systemic treatment.
12. Pregnancy or women of childbearing potential not willing to follow the birth control as described in the informed consent and/or who are breastfeeding.
13. Received unapproved or investigational drug or device within 30 days of the subject's study start date.
14. The judgment of the investigator would make the subject inappropriate for entry into the study.

Device Suizenji (an ultrasound-guided HIFU therapy system) HIFU Treatment Treatment will sonicate at least 50% of the tumor volume. Safety margins between the sonication focus (Red box on the Suizenji screen) to adjacent critical structures such as the bowel and blood vessels will be 10 mm in the anterior-posterior direction and 5 mm in the medial-lateral direction. Subjects will receive the 1st session of HIFU treatment on Day 1. An additional session will be required prior to the initiation of chemotherapy if one of the following; (1) ablation is not completed as planned, or (2) insufficiently ablated per PI's discretion.

If at any time during the treatment procedure, a subject uses the "stop button" indicating pain or discomfort, HIFU treatment will immediately be paused. It will resume only after the subject's pain or discomfort has resolved and the subject is ready to continue. If the subject does not wish to continue on that day, this session can be rescheduled for another day. All HIFU treatment sessions need to be completed prior to the start of chemotherapy.

If any of the following conditions are observed on the day of HIFU treatment, HIFU treatment will be paused until complete resolution:

* Fever exceeding 38°C;
* Impaired consciousness;
* Shock symptoms with systolic blood pressure below 90 mmHg, cold sweat and pallor;
* Jaundice (as judged by the investigators);
* Severe neutropenia, thrombocytopenia, abnormal liver function (increased AST, ALT), abnormal renal function (increased serum creatinine), or increased serum amylase in the most recent clinical examination (severe is defined as Grade 3 or higher in NCI-CTCAE ver. 5.0);
* or any other conditions per investigator's discretion which may not be in the subject's best interest to continue in the study.

If these conditions are not resolved within the HIFU treatment window (prior to initiate the chemotherapy), the subject will be withdrawn the study.

Concomitant and Prohibited medication Standard 1st line chemotherapy FOLFIRINOX (or modified FOLFIRINOX), Gem/nab-PTX, or NALIRIFOX Prohibited previous medications

* Any treatment for pancreatic cancer.
* Investigational medications or investigational medical device within 30 days of the HIFU treatment.

Prohibited concomitant medications (up to 3 months visit)

* Any systemic or local treatment such as immunotherapies, radiotherapy, other adjunctive oncologic treatments to the primary lesion of pancreas as well as to the metastatic lesions.
* Investigational medications or investigational medical device. Safety Assessments Safety and tolerability assessments

  1) Procedure limiting toxicities (up to 30 days post last HIFU treatment)
* Bowel perforation ≥ Grade 3;
* Any other toxicities > Grade 3 with the exception of:

  * Grade 3 abdominal pain unless new and persistent (> 2 weeks duration post HIFU) despite maximal supportive care measures as prescribed by the treating physician;
  * Grade 3 pancreatic duct stenosis, unless new and persistent (> 2 weeks duration post HIFU) despite maximal supportive care measures as prescribed by the treating physician;
  * Grade 3 bile duct stenosis, unless new and persistent (> 2 weeks duration post HIFU) despite maximal supportive care measures as prescribed by the treating physician;
  * Grade 3 fever;
  * Grade 3 pain unless new and persistent (> 2 weeks duration post HIFU) despite maximal supportive care measures as prescribed by the treating physician;
  * Grade 3 increase in lipase or amylase. 2) Adverse events 3) Expected procedure-related local AEs by CTCAE (up to 30 days post last HIFU treatment)
* Pain during and immediately after the HIFU treatment
* Skin redness
* Skin burning 4) Other safety assessments
* Safety lab (hematology, blood chemistry, coagulation, and urinalysis)
* ECG
* Vital Signs/weight
* ECOG-PS
* Numerical Rating Scale (NRS) and analgesics use for abdominal pain Technical Success Assessments In this proposed feasibility study, various options of imaging modalities such as pre- and post-contrast-enhanced CT/MRI, PET-CT and contrast enhanced ultrasonography, and fine needle biopsy will be explored in actual clinical setting (PDAC patients).

Technical success of the HIFU ablation defined as > 50% of treated volume assessed by MRI and/or contrast-enhanced CT after the last HIFU.

In this study, the ablation volume will be assessed post HIFU by the change in volume of hypointensity on non-contrast T1 MRI and by the non-perfused volume (NPV) on contrast-enhanced CT/MRI primary. In addition, other MRI sequences, PET-CT, contrast enhanced ultrasonography, histopathological change data may be collected for exploratory ablation assessment.

Other Assessments Clinical Efficacy Endpoints

* Overall Response Rate up to Month 3 visit
* Change of Tumor volume at primary lesion
* Disease Control Rate
* Tumor Marker (CA19-9, CEA)
* FDG-PET (change from the baseline)
* Immune responses (Tissue, Peripheral blood)
* Numerical Rating Scale (NRS) and analgesics use for abdominal pain
* Long-term oncological outcomes (Progression Free Survival and Overall Survival) Procedure Feasibility Endpoints
* Completion rate of HIFU treatment procedure Study Premature Termination or Study Suspension Criteria If any of the following events occur, the study will be suspended pending DSMB review.
* Any SAE associated with HIFU treatment.
* Any procedure limited toxicities (up to 30 days post last HIFU treatment).
* Any > Grade 3 toxicity associated with HIFU treatment.
* Any death that occurs within 30 days of receiving HIFU treatment.

Either the Sponsor or the PI reserve the right to temporarily suspend or prematurely terminate the study at any time if there is sufficient reasonable cause.

Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to the PI, Sponsor, and FDA.

If the study is prematurely terminated or suspended, the PI will promptly inform the IRB and will provide the reason(s) for the termination or suspension.

Circumstances that may warrant termination or suspension, include, but are not limited to:

* Determination of unexpected, significant, or unacceptable risk to subjects
* Insufficient compliance to protocol requirements
* Data that are not sufficiently complete and/or evaluable The study may resume once concerns about safety, protocol compliance and data quality have been addressed and satisfied by the Sponsor, IRB, and FDA DSMB The membership includes three clinicians (medical oncologist, surgical oncologist, and gastroenterologist) specializing in pancreatic cancer treatment and the medical monitor.

Sample Size Total 10 subjects will be treated.

ELIGIBILITY:
1. Signed an Institutional Review Board (IRB) approved informed consent document.
2. Men and women ≥ 18 years of age.
3. Histologically or cytologically diagnosed PDAC.
4. Newly diagnosed unresectable*, locally advanced or metastatic disease. (* defined as not "Resectable" and not "borderline resectable" based on "Criteria Defining Resectability at Diagnosis" in NCCN Guideline 2024)
5. Primary tumor accessible to HIFU treatment and visualized on transabdominal ultrasonography.
6. Primary tumor site must be a measurable lesion according to RECIST version 1.1 at baseline.
7. ECOG Performance Status (ECOG-PS) of 0 - 1.
8. Life expectancy ≥ 3 months.
9. Adequate organ function defined by:

   * Neutrophil count: ≥ 1,500/mm3
   * Platelet count: ≥ 50,000/mm3
   * Hemoglobin: ≥ 8.0 g/dl
   * Cr: ≤ 1.7 mg/dl
   * AST, ALT: ≤ 3 x upper limit of normal
   * T-Bil: ≤ 2 x upper limit of normal

Exclusion Criteria:

1. Subjects with any cancers other than PDAC who are on active treatment.
2. Subjects who had any prior chemotherapy or interventions for PDAC.
3. Obstructive jaundice (except for subjects who have a bile duct stent placed for obstructive jaundice prior to initiation of HIFU treatment).
4. Tumor embolization in the veins surrounding the pancreas.
5. Cysts outside of primary pancreatic tumor which may obstruct the HIFU sonication pathway. However, if the cyst is completely surrounded by pancreatic tumor, the subject can be included.
6. Subjects with > 50% reduction in caliber of the principal hepatic artery and occlusion of the portal vein seen on preoperative screening CT or MRI scan.
7. Allergy to contrast agents (except when manageable by prophylactic steroid).
8. Subjects having a cardiac pacemaker.
9. Congestive heart failure, symptomatic coronary artery disease, arrhythmia poorly controlled by drugs, history of myocardial infarction or unstable angina within the past 6 months.
10. Subjects with peritoneal dissemination.
11. Active infections requiring systemic treatment.
12. Pregnancy or women of childbearing potential not willing to follow the birth control as described in the informed consent and/or who are breastfeeding.
13. Received unapproved or investigational drug or device within 30 days of the subject's study start date.
14. The judgment of the investigator would make the subject inappropriate for entry into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Technical success for device feasibility | 3 Months
  Technical success of the HIFU ablation defined as > 50% of treated volume assessed by MRI and/or contrast-enhanced CT after the last HIFU. Change from Baseline.

SECONDARY OUTCOMES:
Clinical Efficacy | 3 Months
  Overall Response Rate from baseline up to Month 3 visit
Tumor volume | 3 Months
  Change of Tumor volume at primary lesion from baseline to month 3
Disease Control Rate | 3 months
  Rate of disease spread from baseline to month 3
Tumor Marker | 3 months
  Tumor Marker change from baseline to month 3
FDG-PET | 3 months
  FDG-PET change from the baseline to Month 3
Immune responses | 3 months
  Change from baseline in Immune responses
Numerical Rating Scale (NRS) | 3 months
  Numerical Rating Scale (NRS) and analgesics use for abdominal pain from baseline to Month 3

CONTACTS AND LOCATIONS:
Overall Officials: Pejman Ghanouni, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Increase be treatment options for this patient population